CLINICAL TRIAL: NCT00003531
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Adenocarcinoma of the Pancreas
Brief Title: Antineoplaston Therapy in Treating Patients With Stage IV Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066578; BC-PA-2 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: Adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Stage IV Pancreatic Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Stage IV Pancreatic Cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Stage IV Pancreatic Cancer.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Stage IV Pancreatic Cancer.

DETAILED DESCRIPTION:
Stage IV Pancreatic Cancer patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage IV Pancreatic Cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage IV Pancreatic Cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV adenocarcinoma of the pancreas that is unlikely to respond to existing therapy
* Measurable disease by MRI or CT scan
* Tumor must be at least 2 cm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* No hepatic insufficiency
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* No renal insufficiency
* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No active infection
* No nonmalignant systemic disease
* Not a high medical or psychiatric risk

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy

Surgery:

* Recovered from prior surgery

Other:

* Prior cytodifferentiating agents allowed
* No prior antineoplastons
* No other concurrent antineoplastic agents

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1996-04-10 (Actual); Primary Completion 2005-07-18 (Actual); Study Completion 2005-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with Stage IV Pancreatic Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 15
Completed | 5
Not Completed | 10
Not completed — Not evaluable | 10

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 60.7 [38.6 to 80.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response and Stable Disease
Description: An objective response can be complete or partial. A complete response is complete disappearance of all tumor(s) by physical examination and radiographic studies for a minimum of 4 weeks. A partial response is > 50% reduction in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, lasting for a minimum of four months. Stable disease is < 50% change in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, for a minimum of 12 months.
Time Frame: 14 months
Measure: Number; unit: participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 5
participants
  Stable Disease | 1
  Progressive Disease | 4

ADVERSE EVENTS:
Time Frame: 9 years, 3 months
Description: Fifteen patients were recruited between April 10, 1996 and July 18, 2005. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=15)
Central Venous Catheter Infection (Infections and infestations) | 1
Edema/Fluid retention (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hemorrhage, GI (Gastrointestinal disorders) | 1
Lung (pneumonia) (Infections and infestations) | 2
Confusion (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=15)
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 2
tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Central Venous Catheter Infection (Infections and infestations) | 1
PT (Investigations) | 1
PTT (Investigations) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6
Fever (General disorders) | 1
Rigors/chills (General disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 8
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Gastrointestinal-Other (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Hemorrhage, GI (Gastrointestinal disorders) | 1
Infection (documented clinically): Blood (Infections and infestations) | 1
Lung (pneumonia) (Infections and infestations) | 3
Infection (documented clinically): Mucosa (Infections and infestations) | 1
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Hyperbilirubinemia (Investigations) | 1
Hyperglycemia (Investigations) | 6
Hypernatremia (Investigations) | 8
Hypocalcemia (Investigations) | 2
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 12
Hypomagnesemia (Investigations) | 1
Hyponatremia (Investigations) | 1
SGOT (Investigations) | 4
Confusion (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 2
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 5
Speech impairment (Nervous system disorders) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
Pain: Head/headache (General disorders) | 2
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No